CLINICAL TRIAL: NCT03989622
Title: Evaluation of the Visual Field on the Ground: Impact on Locomotion Rehabilitation Adults With Retinitis Pigmentosa With Loss of Peripheral Vision
Brief Title: Evaluation of the Visual Field on the Ground
Acronym: ECVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I15007
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-04

CONDITIONS: Retinitis Pigmentosa Syndrome
Keywords: Retinitis Pigmentosa
MeSH Terms: conditions — RHYNS syndrome; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evaluation of the visual field on the ground (Experimental): evaluation of the visual field on the ground followed by 10 reeducation sessions
  Interventions: Other: evaluation of the visual field on the ground
- usual care (No Intervention): control session followed by 10 re-education sessions

INTERVENTIONS:
Other: evaluation of the visual field on the ground — evaluation of the visual field on the ground
  Arms: evaluation of the visual field on the ground

SUMMARY:
Retinopathy pigmentosa (which affects about 40,000 patients in France) leads to destruction of the peripheral retina. This condition, often familial, frequently affects young patients. Visual acuity is excellent for a long time, the disease affecting the central macular region only belatedly. On the other hand, the visual field is very quickly narrowed to a central or paracentral zone.

For the patient, knowing the limits of his visual field and learning to adapt is necessary especially when traveling.

The management of these patients is twofold:

* an orthoptist carries out an overall evaluation of the visual field using the Goldmann device (30 cm projection of the areas seen and not seen by the patient's eye), then performs rehabilitation over several weeks
* an instructor of locomotion (open specialization: occupational therapist, case of this project,...) carries out an evaluation in situation, followed by a personalized reeducation over several weeks. The first sessions consist in establishing a climate of confidence, presenting the objectives of the management of locomotion and begin to understand the movements inside and outside accompanied. The following of the rehabilitation is an apprenticeship of the optimal use of the residual field of vision and the proposed technical aids (white cane), in the whole of the displacements, inside and outside.

The residual field of vision is evaluated by a device at the first appointment at the specialized center. This examination, necessary for the professional, is not informative for the patient. It is sometimes supplemented by the evaluation of the visual field of view (ECVS). The ECVS, done jointly by the orthoptist and the locomotion instructor, consists in evaluating the functional visual field on a horizontal plane at 1m (meter) and 5m, and vertical at 5m. The field of vision of the patient, immobile, is materialized by targets deposited at each limit of the zones seen that it indicates.

The investigators believe that the passing of a visual field on the ground, thanks to the projection of the zones of vision, allows the patient to improve his knowledge on his visual possibilities (and gaps) and thus to make his reeducation more efficient.

ELIGIBILITY:
Inclusion Criteria:

* patient at least 18 years old
* patient with retinitis pigmentosa
* a visual field less than or equal to 20 degrees regardless of the degree of visual acuity
* lack of peripheral islets
* to be able to move without a white detection cane
* have signed an informed consent
* be an affiliate or beneficiary of a French social security system.

Exclusion Criteria:

* severe disorders of transparent media that may interfere with visual impairment related to retinitis pigmentosa
* impossibility to follow the protocol
* Limitation of locomotion activities related to other than visual impairments: neurological disorders (hemiplegia, neuropathy, ...)
* musculoskeletal disorders (arthropathies ...)
* Any participation in a protocol having an impact on the walking path by Virtual Reality
* person under the protection of justice, or under guardianship or curators
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
difference in the number of errors committed during a walk between T0 and T2 | 2 months
  difference in the number of errors committed (= number of hurdles, number of "doors" forgotten) during a walk between T0 (before ECVS) and T2 (after ECVS + 10 re-education sessions).

IPD SHARING:
Plan to Share IPD: No